CLINICAL TRIAL: NCT00302315
Title: Effectiveness of Physiotherapy on Postcesarean Pain and Functional Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, İlkim Çıtak Karakaya, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05.T02.102.003
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2006-03

CONDITIONS: Cesarean Section
Keywords: postcesarean physiotherapy; incisional pain; functional activity; connective tissue manipulation; transcutaneous electrical nerve stimulation
MeSH Terms: interventions — Physical Therapy Modalities; Exercise; Transcutaneous Electric Nerve Stimulation; Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Routine care (Active Comparator): All subjects were operated by the same obstetrician (SB) and lower segment transverse incision technique was used for the cesarean section. After delivery, patients were transferred to their rooms within the obstetric ward. Vital signs (heart rate, blood pressure and breathing rate) and body temperatures were assessed regularly. Patients were not allowed to feed orally before bowel movements had started. For post-operative pain control in the first 24 h, meperidine (50 mg, 4 × 1) and non-steroid anti-inflammatory medicine (4 × 1) were administered intravenously. If required by the patient, additional analgesics or anti-inflammatory medications were also administered by the nurses, who were blinded to the group assignment. Patients were encouraged for early ambulation after delivery if they were not hypotensive and uterine bleeding was under control. Initially, they ambulated 10-15 m inside their rooms, and the intensity increased in hours and days. Patients were usually discharged wit
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Thoracic expansion exercises and huffing technique Lower limb exercises TENS with frequency of 120 Hz and pulse width of 60 μs was used for 30 min in every session Connective tissue manipulation (CTM) to the sacral and lumbar regions, Education (proper use of body mechanics during baby caring and daily activities; improving posture; anatomy and functions of the pelvic floor and Knack maneouvre)
  Other Names: exercise; TENS; patient education and recommendations; connective tissue manipulation

SUMMARY:
This study aims to investigate the effectiveness of physiotherapy applications in early postcesarean problems.

DETAILED DESCRIPTION:
This study aims to investigate the effectiveness of physiotherapy applications in early postcesarean problems which make difficulties in functional activities, and includes a physiotherapy intervention group and a control group. Physical characteristics, obstetrical and surgical histories, and systemic problems, back pain, low back pain, headache, urinary/fecal incontinence problems and bowel habit of the subjects both in pregnancy and postpartum periods are recorded. First ambulation time after cesarean, presence of syncope, related vital signs, onset time of bowel peristalsis and defecation are also recorded. Intensities of incisional pain and difficulty in performing functional activities are evaluated by daily 0-10 cm visual analogue scales (VASs). Also, intensities of back pain, low back pain, headache, bloated feeling of the abdomen, and fatigue are also evaluated by daily VASs. Physiotherapy program included breathing exercises, active joint movements of the lower limbs, posture exercises, connective tissue manipulation and transcutaneous electrical nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

cesarean section giving birth to single baby having cesarean under general anesthesia

Exclusion Criteria:

giving birth to multiple babies being followed in intensive care unit after cesarean because of complications

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2004-12; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
incisional pain intensity | Intensity of incision pain was evaluated daily during hospitalization period before the physiotherapy program in the study group.
  Intensity of incision pain was evaluated by horizontal 0-10 cm visual analogue scales (VASs:0 = no pain, 10 = unbearable pain).
intensity of difficulty in functional activities | Intensity of difficulty in functional activities was evaluated daily during hospitalization period before the physiotherapy program in the study group.
  Intensity of difficulty in functional activities was evaluated by horizontal 0-10 cm visual analogue scales (VASs:0 = no difficulty, 10 = unable to perform the activity).
first ambulation time | From transfer to obstetric department room to first ambulation after cesarean
  Time from transfer to obstetric department room to first ambulation after cesarean.
onset time of bowel peristalsis | Only once when breaking gas and defecation occured after Cesarean.
  Time of breaking gas and defecation after Cesarean.

SECONDARY OUTCOMES:
Vital signs | Vital signs were measured before and after first ambulation
  Heart rate, blood pressure, breathing rate and body temperature
Length of staying at the hospital and number of analgesic/anti-inflammatory medication additional to the standard pain control procedure | Only once before discharge from the hospital
  Length of staying at the hospital and number of analgesic/anti-inflammatory medication additional to the standard pain control procedure were recorded, and also cases were observed for any adverse effects which may be due to the physiotherapy applications.

CONTACTS AND LOCATIONS:
Overall Officials: İnci Yüksel, PT. Prof., Study Director — Prof. PT.; İlkim Çıtak Karakaya, PT. PhD., Principal Investigator — Research assistant; Mehmet Gürhan Karakaya, PT. PhD., Study Chair — Research assistant
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)